CLINICAL TRIAL: NCT01241188
Title: A Phase IIb Sensitivity Trial of the Diagnostic Agent C-Tb, When Given Intradermally by the Mantoux Technique to Adult Patients Recently Diagnosed With Active TB
Brief Title: A Trial of the C-Tb Skin Test, When Given Intradermally to Adult Patients Recently Diagnosed With Active Tuberculosis (TB)
Acronym: TESEC-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-04
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
Keywords: tuberculosis; rdESAT-6; CFP-10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1 µg/0.1 mL C-Tb (Experimental): The C-Tb and 2 TU Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: C-Tb
- 2 TU Tuberculin PPD RT 23 SSI (Active Comparator): The C-Tb and 2 TU Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: 2 TU Tuberculin PPD RT 23 SSI

INTERVENTIONS:
Biological: C-Tb — The C-Tb agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearms according to a double blind randomisation scheme
  Other Names: rdESAT-6 + rCFP-10
  Arms: 0.1 µg/0.1 mL C-Tb
Biological: 2 TU Tuberculin PPD RT 23 SSI — The 2 TU Tuberculin PPD RT 23 SSI agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearms according to a double blind randomisation scheme
  Other Names: PPD; Tuberculin
  Arms: 2 TU Tuberculin PPD RT 23 SSI

SUMMARY:
Tuberculosis (TB) continues to be the most important bacterial infection worldwide and therefore new improved diagnostic tests are needed to help doctors in diagnosing TB.

The new skin test is named C-Tb. Like the current Tuberculin Skin Test (TST), the C-Tb test is injected just under the skin and will when positive show a redness and/or swelling at the injection site while a negative test will leave no reactions.

The aim of this trial is to test the C-Tb skin test in adults diagnosed with TB to determine if a TB infected individual has a truly positive test result (this is called to find the sensitivity of the skin test).

DETAILED DESCRIPTION:
The trial is designed to investigate the sensitivity of C-Tb using various sizes of cut-off of induration in a double blind randomised, split-body study comparing 0.1 µg/0.1 mL C-Tb with the reference agent 2 T.U. Tuberculin PPD RT23 SSI. (Each volunteer receives the C-Tb agent in one arm and 2 T.U. Tuberculin PPD RT 23 SSI in the other arm). Two groups of adult patients recently diagnosed with active TB will be investigated; patients in the main group will NOT have a co-infection with HIV and patients in the second group will have a co-infection with HIV.

The C-Tb and 2 TU Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a double blind randomisation scheme.

The primary objectives are to assess the sensitivity of the C-Tb test as a function of the cut-off value (i.e., the smallest size of induration measured in mm resulting in a positive outcome of the C-Tb test) when the test is administered intradermally by the Mantoux technique to HIV negative adult patients recently diagnosed with active TB and to assess the sensitivity of the C-Tb test as a function of the cut-off value (i.e., the smallest size of induration measured in mm resulting in a positive outcome of the C-Tb test) when the test is administered intradermally by the Mantoux technique to HIV positive adult patients recently diagnosed with active TB The sensitivity is defined as the relative frequency of patients with an induration response ≥ cut-off in TB patients.

Similarly the specificity of the C-Tb test is defined as the relative frequency of subjects in a healthy population (i.e., no exposure to M. tuberculosis) who have an induration response < cut-off after a C-Tb test.

An optimal cut-off point of being infected will be determined by combing the results from the present sensitivity study with those from a parallel specificity study in (BCG vaccinated) individuals with no previous exposure to M. tuberculosis.

The secondary objectives of the trial is to compare the induration response of C-Tb with the induration response of 2 T.U. Tuberculin PPD RT 23 SSI, to compare the induration response of C-Tb with the in-vitro IFN-γ response measured at screening using the QuantiFERON®-TB Gold In Tube assay, to correlate the induration response to the initial CD4+ counts in HIV positive patients and to record all adverse events (local and systemic) occurring within 28 days after application of the agents

ELIGIBILITY:
Inclusion Criteria (HIV negative patients):

1. Has signed an informed consent
2. Aged 18 to 65 years
3. Has been diagnosed with active TB:

   1. has a compatible clinical picture of TB according to South African guidelines with the intention to treat and at least 1 documented positive sputum smear microscopy result or
   2. has a compatible clinical picture of TB according to South African Guidelines with the intention to treat and a positive culture result
4. Is HIV negative confirmed by 2 two rapid tests (Abbott-DetermineTM HIV-1/2 and Sensa (Seyama Solutions, SA))
5. Is willing and likely to comply with the trial procedures
6. Is prepared to grant authorized persons access to their medical record

Inclusion Criteria (HIV positive patients):

1. Has signed an informed consent
2. Aged 18 to 65 years
3. Has a compatible clinical picture of TB according to South African guidelines with the intention to treat
4. Is HIV positive confirmed by:

   1. 2 positive rapid tests (Abbott-DetermineTM HIV-1/2 and Sensa (Seyama Solutions, SA)) or
   2. 1 positive rapid tests (Abbott-DetermineTM HIV-1/2 or Sensa (Seyama Solutions, SA)) and an additional confirmatory ELISA (Enzygnost anti-HIV-1/2 Plus)
5. Is willing and likely to comply with the trial procedures
6. Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

1. Has been in treatment for TB for more than 2 weeks
2. Has a known MDR/XDR-TB
3. Has within 3 months prior to the day of inclusion been in treatment with a product which is likely to modify the immune response except for HIV treatment (e.g., immunoglobulin, systemic corticosteroids, methotrexate, azathioprine, cyclosporine or blood products)
4. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines)
5. Has been vaccinated with BCG < 6 months prior to the day of inclusion
6. Has been tuberculin (TST) tested < 6 months prior to the day of inclusion
7. Has an active disease affecting the lymphoid organs except for HIV (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
8. Has a current skin condition which interferes with the reading of the skin tests e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
9. Has a condition where blood drawings pose more than minimal risk for the patient, such as haemophilia, other coagulation disorders, or significantly impaired venous access
10. Currently participating in another clinical trial with an investigational or non investigational drug or device, or has participated in another clinical trial within the 3 months prior to dosing
11. Has participated in previous clinical trials investigating the ESAT-6 and/or CFP-10 antigens
12. Is pregnant, breastfeeding or intending to get pregnant
13. Has a condition which in the opinion of the investigator is not suitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The diameter of induration at the injection sites measured transversely to the long axis of the forearm 2-3 days after application of the agents | From injections to 2-3 days after aplication

SECONDARY OUTCOMES:
Injection site adverse reactions within 28 days after application of the agents | Onset between the injections and 28 days after the injections
All adverse events occurring within 28 days after application of the agents | Onset between the injections and 28 days after the injections
Laboratory safety parameters of haematology and biochemistry | Onset between the injections and 28 days after the injections
In vitro IFN-γ response as measured by the QuantiFERON®-TB Gold In Tube assay | Onset between the injections and 28 days after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Thierry-Carstensen, Study Director — Statens Serum Institut Denmark; Keertan Dheda, MD, Principal Investigator — University of Cape Town Lung Institute (Pty) Ltd, South Africa
Locations (1):
- University of Cape Town Lung Institute (Pty) Ltd, Cape Town, Cape Town, South Africa

REFERENCES:
- [Derived] Hoff ST, Peter JG, Theron G, Pascoe M, Tingskov PN, Aggerbeck H, Kolbus D, Ruhwald M, Andersen P, Dheda K. Sensitivity of C-Tb: a novel RD-1-specific skin test for the diagnosis of tuberculosis infection. Eur Respir J. 2016 Mar;47(3):919-28. doi: 10.1183/13993003.01464-2015. Epub 2015 Dec 17. PMID 26677940
- [Derived] Aggerbeck H, Giemza R, Joshi P, Tingskov PN, Hoff ST, Boyle J, Andersen P, Lewis DJ. Randomised clinical trial investigating the specificity of a novel skin test (C-Tb) for diagnosis of M. tuberculosis infection. PLoS One. 2013 May 14;8(5):e64215. doi: 10.1371/journal.pone.0064215. Print 2013. PMID 23691171